CLINICAL TRIAL: NCT04180748
Title: Survey of Diversity and Density on the Facial Bacteriome of Different Skin Types
Brief Title: Survey of the Facial Bacteriome
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5749
Record Dates: First submitted 2019-11-21; First posted 2019-11-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Understanding Skin Health and the Microbiome; Microbial Colonization
Keywords: Microbiome; Dermatology; Cosmetics; Autofluorescence
MeSH Terms: conditions — Communicable Diseases | interventions — Optical Imaging; Light

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal skin
  Interventions: Other: fluorescence imaging with 405nm light
- Oily skin
  Interventions: Other: fluorescence imaging with 405nm light
- Dry skin
  Interventions: Other: fluorescence imaging with 405nm light
- Combination skin
  Interventions: Other: fluorescence imaging with 405nm light
- Sensitive skin
  Interventions: Other: fluorescence imaging with 405nm light

INTERVENTIONS:
Other: fluorescence imaging with 405nm light — Each group will have images taken with an Health Canada approved device to capture images under white light and 405nm fluorescence with an mCherry filter. These images will not be used for diagnostics and will be analyzed for features which correlate to identified microbes from 16S RNA analysis and traditional microbiological technique. Groups are self identified by participants in order to capture a diverse population.

SUMMARY:
The microbiome can affect skin health from the gut-skin axis, from environmental exposure, and topical treatments. Decreasing biodiversity of skin microbiota has been linked to inflammatory conditions, allergies, and skin health.

This cross sectional study will be used to survey healthy volunteers and measure the density and diversity of skin flora of varying skin types. The aim of this study is to identify associations between the skin flora and characteristics of healthy skin types.

DETAILED DESCRIPTION:
The microbiome can affect skin health from the gut-skin axis, from environmental exposure, and topical treatments. Decreasing biodiversity of skin microbiota has been linked to inflammatory conditions, allergies and skin health.

Therefore, this cross sectional study will be used to survey healthy volunteers and measure the density and diversity of skin flora of varying skin types.

This study will aim to determine if there are associations between the diversity and/or density of normal bacterial flora and (1) the different skin types (i.e. normal, dry, oily, combination, sensitive); (2) the different Fitzpatrick skin types (i.e. ivory; fair or pale; fair to beige with golden undertones; olive or light brown; dark brown; deeply pigmented dark brown to darkest brown): (3) the number of skin products used daily representing time spent on skin health (i.e. low:0-1, mid:2-4, high:5+). Participants will complete a survey in which they will identify their skin conditions and the number and type of skin products they use on their face as a part of their daily routine.

In addition, this study will evaluate the potential of an autofluorescence image-guided device to capture differences in healthy human skin flora through autofluorescence. The MolecuLight i:X™ is used to detect bacteria in chronic wounds. Based on extensive preclinical and clinical studies, the i:X has demonstrated its capability at collecting autofluorescent images of wounds and detecting the presence and relative changes in connective tissue (e.g. collagen) content and bio-distribution involved in wound healing. It can also detect the presence and relative amounts of commensal and pathogenic bacteria within the wound based on autofluorescence alone (these bacteria are invisible to standard visualization with the naked eye using white light), thus providing a measure of infection status.

The imaging device will be used to image skin from the cheek and forehead of healthy volunteers to compare the fluorescent characteristics of normal skin flora. The fluorescent images captured with the i:X™ will be compared against 16S RNA analysis of the skin microbiome and traditional microbiology techniques with selective and differential tests. In addition, non-selective agars will be used to grow bacteria according to the spatial topography of the skin, using a tape stripping method, with lightly adhesive 3M™Tegaderm wound dressings. This will serve as a "map" for fluorescent images by which to compare fluorescent features to bacterial species.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 18 years or older.
* Able to provide consent
* Identifies as having normal (n=6), oily (n=6), dry (n=6), combination (n=6), and/or sensitive (n=6) skin groups.

Exclusion Criteria:

* Treatment with topical or oral antibiotic(s) or antifungal(s) within 1 month of enrolment
* Diagnosed with chronic conditions (excluding acne and dermatological conditions)
* Treatment for a chronic condition
* Diagnosed with bacterial/fungal infection within 1 month of enrolment
* Treatment with an investigational drug within 1 month of enrolment
* Allergies to antibiotics, antiseptics, tape, or adhesives
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy volunteers with no existing or recent skin conditions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Bacterial diversity between individuals of each skin condition (i.e. normal, dry, oily, combination, sensitive). (Number of CFU) | February 2020
  Frequency of unique colonies identified from microbiological and microbiome techniques between individuals of each skin condition (i.e. normal, dry, oily, combination, sensitive).
Bacterial density (CFU/cm2) between individuals of each skin condition | February 2020
  Abundance of bacterial colonies per cm2 of sampled area identified from microbiological and microbiome techniques between individuals of each skin condition (i.e. normal, dry, oily, combination, sensitive).
MolecuLight i:X detection of density and diversity (green or red fluroescence/cm2) | February 2020
  Abundance of green and/or red fluorescent detection with MolecuLight i:X per cm2 of sampled area between individuals of each skin condition. Frequency of green or red fluorescence per sample.

SECONDARY OUTCOMES:
Identification of spatial distribution of bacterial species (CFU/cm2 of individual species) | February 2020
  Abundance of unique species and bacterial families identified from microbiological and microbiome techniques between individuals of each skin condition (i.e. normal, dry, oily, combination, sensitive) and Fitzpatrick skin type per. Distribution of unique species and bacterial families across the area of sampling of individuals on Tegaderm "map".
Identification of spatial distribution of red/green fluorescence detected with MolecuLight i:X™ (red and green fluroescence/cm2) | February 2020
  Abundance of unique fluorescent (green and red) detection with MolecuLight i:X™ between individuals of each skin condition (i.e. normal, dry, oily, combination, sensitive) and Fitzpatrick skin type. Distribution of red and green fluorescent signals across the area of sampling of individuals on Tegaderm "map".

OTHER OUTCOMES:
Imapact of cosmetic use on diversity of bacterial species across individuals with different cosmetic use (high, mid, low). (Number of CFU) | February 2020
  Compare the frequency of specific bacterial species and bacterial families identified with microbiology and microbiome techniques between individuals with different skin care routines.
Imapact of cosmetic use on density of bacterial species across individuals with different cosmetic use (high, mid, low). (CFU/cm2) | February 2020
  Compare the abundance of specific bacterial species and bacterial families identified with microbiology and microbiome techniques between individuals with different skin care routines per cm2 of area sampled.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Research Tower, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD which underlie results may be shared in an academic publication. It is undecided if these results may yield a publication.

REFERENCES:
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Luckey TD. Introduction to intestinal microecology. Am J Clin Nutr. 1972 Dec;25(12):1292-4. doi: 10.1093/ajcn/25.12.1292. No abstract available. PMID 4639749
- [Background] Sender R, Fuchs S, Milo R. Revised Estimates for the Number of Human and Bacteria Cells in the Body. PLoS Biol. 2016 Aug 19;14(8):e1002533. doi: 10.1371/journal.pbio.1002533. eCollection 2016 Aug. PMID 27541692
- [Background] Burne RA, Quivey RG Jr, Marquis RE. Physiologic homeostasis and stress responses in oral biofilms. Methods Enzymol. 1999;310:441-60. doi: 10.1016/s0076-6879(99)10035-1. PMID 10547811
- [Background] Robinson CJ, Bohannan BJ, Young VB. From structure to function: the ecology of host-associated microbial communities. Microbiol Mol Biol Rev. 2010 Sep;74(3):453-76. doi: 10.1128/MMBR.00014-10. PMID 20805407
- [Background] Davey ME, O'toole GA. Microbial biofilms: from ecology to molecular genetics. Microbiol Mol Biol Rev. 2000 Dec;64(4):847-67. doi: 10.1128/MMBR.64.4.847-867.2000. PMID 11104821
- [Background] Salem I, Ramser A, Isham N, Ghannoum MA. The Gut Microbiome as a Major Regulator of the Gut-Skin Axis. Front Microbiol. 2018 Jul 10;9:1459. doi: 10.3389/fmicb.2018.01459. eCollection 2018. PMID 30042740
- [Background] Prescott SL, Larcombe DL, Logan AC, West C, Burks W, Caraballo L, Levin M, Etten EV, Horwitz P, Kozyrskyj A, Campbell DE. The skin microbiome: impact of modern environments on skin ecology, barrier integrity, and systemic immune programming. World Allergy Organ J. 2017 Aug 22;10(1):29. doi: 10.1186/s40413-017-0160-5. eCollection 2017. PMID 28855974
- [Background] Lee HJ, Jeong SE, Lee S, Kim S, Han H, Jeon CO. Effects of cosmetics on the skin microbiome of facial cheeks with different hydration levels. Microbiologyopen. 2018 Apr;7(2):e00557. doi: 10.1002/mbo3.557. Epub 2017 Nov 29. PMID 29193830
- [Background] Sohn E. Skin microbiota's community effort. Nature. 2018 Nov;563(7732):S91-S93. doi: 10.1038/d41586-018-07432-8. No abstract available. PMID 30464283
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Stone FM, Coulter CB. PORPHYRIN COMPOUNDS DERIVED FROM BACTERIA. J Gen Physiol. 1932 Jul 20;15(6):629-39. doi: 10.1085/jgp.15.6.629. PMID 19872672
- [Background] Philipp-Dormston WK, Doss M. Comparison of porphyrin and heme biosynthesis in various heterotrophic bacteria. Enzyme. 1973;16(1):57-64. doi: 10.1159/000459362. No abstract available. PMID 4208581
- [Background] Kjeldstad B, Christensen T, Johnsson A. Porphyrin photosensitization of bacteria. Adv Exp Med Biol. 1985;193:155-9. doi: 10.1007/978-1-4613-2165-1_18. No abstract available. PMID 4096295
- [Background] Cox CD, Adams P. Siderophore activity of pyoverdin for Pseudomonas aeruginosa. Infect Immun. 1985 Apr;48(1):130-8. doi: 10.1128/iai.48.1.130-138.1985. PMID 3156815
- [Background] Cody YS, Gross DC. Characterization of Pyoverdin(pss), the Fluorescent Siderophore Produced by Pseudomonas syringae pv. syringae. Appl Environ Microbiol. 1987 May;53(5):928-34. doi: 10.1128/aem.53.5.928-934.1987. PMID 16347352
- [Background] Agren MS, Werthen M. The extracellular matrix in wound healing: a closer look at therapeutics for chronic wounds. Int J Low Extrem Wounds. 2007 Jun;6(2):82-97. doi: 10.1177/1534734607301394. PMID 17558006
- [Background] DaCosta RS, Kulbatski I, Lindvere-Teene L, Starr D, Blackmore K, Silver JI, Opoku J, Wu YC, Medeiros PJ, Xu W, Xu L, Wilson BC, Rosen C, Linden R. Point-of-care autofluorescence imaging for real-time sampling and treatment guidance of bioburden in chronic wounds: first-in-human results. PLoS One. 2015 Mar 19;10(3):e0116623. doi: 10.1371/journal.pone.0116623. eCollection 2015. PMID 25790480
- [Background] Wu YC, Kulbatski I, Medeiros PJ, Maeda A, Bu J, Xu L, Chen Y, DaCosta RS. Autofluorescence imaging device for real-time detection and tracking of pathogenic bacteria in a mouse skin wound model: preclinical feasibility studies. J Biomed Opt. 2014 Aug;19(8):085002. doi: 10.1117/1.JBO.19.8.085002. PMID 25089944
- [Background] He SY, McCulloch CE, Boscardin WJ, Chren MM, Linos E, Arron ST. Self-reported pigmentary phenotypes and race are significant but incomplete predictors of Fitzpatrick skin phototype in an ethnically diverse population. J Am Acad Dermatol. 2014 Oct;71(4):731-7. doi: 10.1016/j.jaad.2014.05.023. Epub 2014 Jun 11. PMID 24928709
- [Background] Baumann L. Understanding and treating various skin types: the Baumann Skin Type Indicator. Dermatol Clin. 2008 Jul;26(3):359-73, vi. doi: 10.1016/j.det.2008.03.007. PMID 18555952
- [Background] Ottolino-Perry K, Chamma E, Blackmore KM, Lindvere-Teene L, Starr D, Tapang K, Rosen CF, Pitcher B, Panzarella T, Linden R, DaCosta RS. Improved detection of clinically relevant wound bacteria using autofluorescence image-guided sampling in diabetic foot ulcers. Int Wound J. 2017 Oct;14(5):833-841. doi: 10.1111/iwj.12717. Epub 2017 Feb 28. PMID 28244218
- [Background] Chamma E, Qiu J, Lindvere-Teene L, Blackmore KM, Majeed S, Weersink R, Dickie CI, Griffin AM, Wunder JS, Ferguson PC, DaCosta RS. Optically-tracked handheld fluorescence imaging platform for monitoring skin response in the management of soft tissue sarcoma. J Biomed Opt. 2015 Jul;20(7):076011. doi: 10.1117/1.JBO.20.7.076011. PMID 26214616
- [Background] Wu YC, Smith M, Chu A, Lindvere-Teene L, Starr D, Tapang K, Shekhman R, Wong O, Linden R, DaCosta RS. Handheld fluorescence imaging device detects subclinical wound infection in an asymptomatic patient with chronic diabetic foot ulcer: a case report. Int Wound J. 2016 Aug;13(4):449-53. doi: 10.1111/iwj.12451. Epub 2015 Apr 22. PMID 25907362
- See also: Understanding Your Skin. Different skin conditions as defined by cosmetic industry — http://www.en.eucerin.ca/about-skin/basic-skin-knowledge/skin-types.